CLINICAL TRIAL: NCT03159325
Title: Delivery of Self-management Through a Peer-support Telehealth Intervention in Patients With Cardiovascular Disease: The Healing Circles Project
Brief Title: The Healing Circles Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Scott Lear, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H16-03203
Record Dates: First submitted 2017-05-03; First posted 2017-05-18 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Heart Diseases; Cardiovascular Diseases
Keywords: internet; chronic disease management; technology; telehealth; application
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The usual care group will receive all standard treatment, instructions and information for patients with cardiovascular disease, but no Healing Circles program.
- Healing Circles (Experimental): Healing Circles is an evidence-based and patient-informed novel self-management platform designed to support patients with CVD. It uses a private, secure social network that helps connect patients to one another, to personalized, disease management information , and provides functions to assist patients in self-management via evidence-based principles of behaviour change.
  Interventions: Behavioral: Healing Circles

INTERVENTIONS:
Behavioral: Healing Circles — See description in the arm description.
  Arms: Healing Circles

SUMMARY:
Heart disease is a leading cause of death and disability in Canada. Providing social and peer supports has been proven to help patients manage their health and stay out of the hospital. The use of telehealth has opened up a wider possibility of patients receiving peer support while staying in their homes and communities. The investigators plan to study a new application for supporting patients through peer support. The application can be accessed by smartphone, tablet and desktop/laptop computer. Over two years, the investigators anticipate that the application (Healing Circles) will improve patient self care and reduce hospitalizations.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of death and disability in Canada costing $22.2 billion annually in health care costs and lost productivity. Cardiovascular diseases are complex conditions that afflict older adults more so than any other population. As CVD is a chronic condition, many patients live with their disease and are affected by it on a daily basis in their homes and communities. Unfortunately, many patients 'suffer' in isolation. It is well-accepted that patient self-management plays a key role in improving patient health and reducing hospital admissions. Social and peer support, as well as timely access to credible information on managing CVD are essential for patient self-management.

While there is a growing understanding that patients with CVD benefit from being actively engaged in their own care, questions remain as to where and how self management support should be delivered. Integration of self-management programs within the health care system has been a challenge due to the system emphasis on the management of acute and episodic conditions rather than the less intense and more drawn-out patient interactions characteristic of chronic conditions. Clearly alternatives are needed to support patient self-management and reduce needless hospital admissions.

The rise in technology and telecommunications has opened up an array of possibilities for patients to be connected to their health while remaining in their homes and community. Outside of the health care sector, peer support and social networking have seen tremendous growth through the use of telecommunications. The value of these networks to improving health and self-management, however, has not been robustly studied.

Through an existing partnership between university-based researchers, industry (Curatio), decision-makers (Vancouver Coastal Health), clinicians and patients the investigators have developed a peer support and self-management platform called Healing Circles. The investigator's 10-week pilot study of Healing Circles in patients with ischemic heart disease demonstrated the feasibility and acceptability, and resulted in key improvements to social support and self-management, as well as demonstrated ease of use of the application itself. The current proposal represents the next phase in our program to scale-up and spread the use of Healing Circles.

The primary hypothesis is that patients with CVD using the Healing Circles platform will have improved self-management skills compared to patients receiving usual care. Secondary hypotheses are that participation in Healing Circles application will improve quality of life and health service use (and associated costs). Outcomes of end-user perceptions, attitudes and satisfaction with the platform will also be assessed.

Participants (n=250) will be recruited through cardiology and cardiac outpatient clinics in Greater Vancouver, as well as through community presentations and mailouts. Patients with documented CVD, who have regular access to a device that supports Healing Circles (computer, tablet or smartphone) will be randomized to either the Healing Circles application or usual care and followed for up to a 2.5 year period.

Healing Circles participants will form 'Circles' with 8 to 10 other participants to connect with and support one another as they learn to live day-to-day with their CVD. Patients also have the ability to connect and engage all members of the wider Healing Circles community. The investigators anticipate that participation in Healing Circles will support patient self-management for patients in their homes resulting in reduced need for health care and hospital use.

ELIGIBILITY:
Inclusion Criteria:

(i) men and women with CVD (ischemic heart disease, atrial fibrillation, heart failure and patients with implantable cardioverter-defibrillator); (ii) at least 18 years of age; (iii) own, or have regular access to, either a smartphone (Android or iOS operating system), tablet or laptop/desktop computer; and (iv) able to understand English.

Exclusion Criteria:

(i) patients with planned surgical intervention (will be approached after surgery); (ii) another household member in the study; and (iii) unable to provide informed consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in patient self-management (Health Education Impact Questionnaire v3.0) every 6 months until study end. | At baseline (0 years) and followed for 2.5 years, for a total of 2 to 6 assessments per subject
  In this 40 item questionnaire, participants will be asked to answer questions related to life engagement, health behaviours, skill acquisition, constructive attitudes, self-monitoring, health service navigation, social support, and emotional well-being.

SECONDARY OUTCOMES:
Health-related Quality of Life (EuroQol 5D5L) | At baseline (0 years) and followed for 2.5 years, for a total of 2 to 6 assessments per subject
  In this 5-item questionnaire, participants will be asked to answer questions related to mobility, self-care, your usual activities, pain/discomfort, anxiety/depression.
Subjective Quality of Life (ICECAP-A) | At baseline (0 years) and followed for 2.5 years, for a total of 2 to 6 assessments per subject
  In this 5-item questionnaire, participants will be asked to answer questions related to feeling settled and secure, love and friendship, independence, achievements, enjoyment and pleasure.
Health Resource Use (study specific questionnaire) | At baseline (0 years) and followed for 2.5 years, for a total of 2 to 6 assessments per subject
  In this questionnaire, participants will be asked to answer questions about the heath services you have used in the past six months (e.g., health professional visits, hospitalizations, medication use, as well as work and time off of work due to health issues).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lear, PhD, Principal Investigator — Simon Fraser University; Brodie Sakakibara, PhD, Study Director — University of British Columbia
Locations (4):
- Canada (4):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Northern Health Authority, Prince George, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakakibara BM, Chakrabarti S, Krahn A, Mackay MH, Sedlak T, Singer J, Whitehurst DG, Lear SA. Delivery of Peer Support Through a Self-Management mHealth Intervention (Healing Circles) in Patients With Cardiovascular Disease: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 11;8(1):e12322. doi: 10.2196/12322. PMID 30635261